CLINICAL TRIAL: NCT07050641
Title: An Open Multi-center Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of SCTB39-1 in Adult Patients With Advanced Malignant Solid Tumours
Brief Title: Phase I/II Study of SCTB39-1 in Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCTB39-1-X201
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Advanced Malignant Solid Tumor
Keywords: advanced malignant solid tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCTB39-1 (Experimental): SCTB39-1 of different doses, IV, every 3 weeks
  Interventions: Drug: SCTB39-1

INTERVENTIONS:
Drug: SCTB39-1 — SCTB39-1, IV

SUMMARY:
This study aims to evaluate the safety, tolerability, PK characteristics, immunogenicity, and preliminary anti-tumor efficacy of SCTB39-1 as a monotherapy in adult patients with advanced malignant solid tumours. This study is an open label, multicentre, dose-escalation and dose-expansion Phase I/II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form (ICF);
2. Male or female, over 18 years old;
3. Survival duration more than 3 months;
4. ECOG score ≤ 1 point;
5. Participants in Phase Ia (dose-escalation phase) are required to meet the following criteria: histologically or cytologically confirmed diagnosis of advanced malignant solid tumour;
6. Participants in Phase Ib (dose-expansion phase) and Phase II are required to meet the following criteria: Histologically or cytologically confirmed specific type advanced malignant solid tumours;
7. At least one measurable tumor lession according to RECIST v1.1;
8. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Has participated in another clinical study within 4 weeks prior to the first dose;
2. Other malignancies diagnosed within 5 years prior to the enrollment;
3. Participants with brainstem, meningeal, spinal metastases, or compression; active central nervous system metastases;
4. Significant bleeding risk;
5. Presence of pleural effusion, peritoneal effusion, or ascites;
6. History of permanent discontinuation of immunotherapy due to immune-related toxicity or occurrence of ≥ Grade 3 irAEs;
7. Presence of any active autoimmune disease or a history of autoimmune disease with an expected recurrence;
8. History of severe allergies, severe drug allergies (including unapproved investigational drugs);
9. History of organ transplantation or stem cell transplantation;
10. Need for immunosuppressive drugs within 2 weeks prior to enrollment or anticipated during the study;
11. Received chemotherapy, immunotherapy, biologic therapy, or other anti-tumor treatments within 4 weeks before enrollment;
12. Pregnant or breastfeeding female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting toxicity(DLT) | From Day 0 up to Day 21
  Incidence of dose-limiting toxicities up to the Day 21 visit
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD based on RECIST Version 1.1.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with SCTB39-1 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment with SCTB39-1 until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Science, Beijing, China

IPD SHARING:
Plan to Share IPD: No